CLINICAL TRIAL: NCT02847533
Title: Inflammatory Markers and Resistant Depression
Acronym: InDep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: API/2014/50
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Depression
Keywords: resistant depression; inflammation
MeSH Terms: conditions — Depression; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- resistant depression (Other): patients suffering from resistant unipolar depression (at least 2 failed antidepressant treatments for the current episode)
  Interventions: Procedure: blood sample; Behavioral: psychometric scales
- non resistant depression (Other): patients in remission from unipolar depressive disorder
  Interventions: Procedure: blood sample; Behavioral: psychometric scales

INTERVENTIONS:
Procedure: blood sample — blood sample for concentration levels of inflammatory markers
Behavioral: psychometric scales — Mini international interview MADRS, C-SSRS, QIDS-SR, BIS-10, BDHI, BART, ERD

SUMMARY:
This study focuses on blood inflammatory markers (pro-inflammatory cytokines, anti-inflammatory cytokines, monocytes costimulation molecules) in patients with resistant unipolar depression in comparison with non-resistant unipolar depressed patients.

ELIGIBILITY:
Inclusion Criteria:

* group 1: Patients with resistant MDD (at least 2 failed treatments for the current episode) ,current treatment with IRS or IRSNA,
* group 2: patients with MDD remission after response to an antidepressant treatment.

Exclusion Criteria:

* comorbid somatic or psychiatric disorders: chronic or acute inflammatory diseases, previous treatment with brain stimulation for the current episode, legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
plasmatic concentration of Interleukin 6 | at patient inclusion

SECONDARY OUTCOMES:
concentration of proinflammatory cytokine | at patient inclusion
  Expression intensity of monocytes costimulation molecules
concentration of antiinflammatory cytokine | at patient inclusion
functional polymorphisms of expression genes of inflammatory proteins | at patient inclusion
plasmatic concentration of Retinoid X receptor signaling pathway | at patient inclusion
Expression rate of monocytes costimulation molecules | at patient inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Haffen, MD PhD, Principal Investigator — CHU Besançon
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided